CLINICAL TRIAL: NCT00621491
Title: Randomized Controlled Clinical Trial for Prevention of Thromboembolic Complications After Permanent Transvenous Leads Implantation in High-risk Patients
Brief Title: Prevention of Venous Thrombosis After Permanent Transvenous Leads Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Roberto Costa, MD PhD, Associate Professor of Cardiovascular Surgery, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SDC 2273/03/067
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2008-01

CONDITIONS: Cardiac Pacing; Complications; Venous Thrombosis
Keywords: cardiac pacing; pacing complication; venous thrombosis; warfarin; anticoagulation; randomized trial
MeSH Terms: conditions — Venous Thrombosis | interventions — Warfarin; Anticoagulants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator): Single daily dose of Placebo during six months
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Single daily dose of Warfarin (5 mg/orally), adjusted to achieve an International Normalized Ratio (INR) between 2 to 3.5 times the normal value during six months
  Other Names: oral anticoagulants

SUMMARY:
The aim of this study was to compare the safety and efficacy of warfarin versus placebo, administered for 6 months, in the prevention of thromboembolic complications after transvenous cardiac devices implantation in high-risk patients.

DETAILED DESCRIPTION:
Venous lesions following cardiac devices implantation are a common complication of transvenous access that may cause disease manifestations and difficulties during reoperations. These lesions tend to develop early, and their incidence decreases gradually within 6 months after device implantation. Ventricular dysfunction and previous transvenous temporary leads ipsilateral to the permanent implant are risk factors identified in a previous study performed at our institution and other risk factors have been reported recently.The usefulness of prophylactic therapeutic strategies to prevent these complications, however,remains unknown. This randomized trial examined the effects of warfarin in the prevention of these complications in high-risk patients. After device implantation, patients were randomly assigned to receive either placebo or warfarin. Periodical clinical and laboratorial evaluations were performed to anticoagulant management. Following the six-month period, every patient was submitted to a digital subtraction venography.

ELIGIBILITY:
Inclusion Criteria:

* adults patients submitted to first transvenous implant of pacemakers, implantable cardioverter-defibrillator, or cardiac resynchronization therapy devices
* left ventricular ejection fraction ≤0.40 and/or
* previous transvenous temporary leads ipsilateral to the permanent device implant

Exclusion Criteria:

* history of venous thromboembolism
* atrial fibrillation
* coagulopathy or platelet disorder
* malignancy
* gastro-intestinal hemorrhage or active gastro-duodenal ulcer in the past 6 months
* abnormal prothrombin time (PT)or an international normalized ratio (INR) >40%, or treated with oral anticoagulants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of venous obstructions observed by digital subtraction venography | Six months

SECONDARY OUTCOMES:
Safety of anticoagulant therapy, morbidity and overall mortality | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Costa, MD PhD, Study Chair — University of Sao Paulo; Katia R Silva, RN PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute (InCor) - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Costa R, Da Silva KR, Rached R, Martinelli Filho M, Carnevale FC, Moreira LF, Stolf NA. Prevention of venous thrombosis by warfarin after permanent transvenous leads implantation in high-risk patients. Pacing Clin Electrophysiol. 2009 Mar;32 Suppl 1:S247-51. doi: 10.1111/j.1540-8159.2008.02295.x. PMID 19250106
- [Result] Silva KR, Costa R, Abi Rached R, Martinelli Filho M, Caldas JG, Carnevale FC, Moreira LF, Stolf NA. Warfarin prevents venous obstruction after cardiac devices implantation in high-risk patients: partial analysis. Rev Bras Cir Cardiovasc. 2008 Oct-Dec;23(4):542-9. doi: 10.1590/s0102-76382008000400015. English, Portuguese. PMID 19229428